CLINICAL TRIAL: NCT05461950
Title: Feasibility-testing of Extra-uterine Placental Transfusion to Facilitate Intact-cord Stabilisation and Physiology-based Cord Clamping for Term and Preterm Infants Delivered by Acute or Planned Caesarean Section
Brief Title: Intact-cord Stabilisation and Physiology-based Cord Clamping in Caesarean Sections
Acronym: INTACT
Status: Completed | Type: Observational
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 399101
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Cesarean Section; Infant Conditions
Keywords: infant stabilisation; intact umbilical cord; umbilical cord clamping; placental transfusion; cesarean section
MeSH Terms: conditions — Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Self-breathing infants: Vigorous infants with spontaneous onset of respiration within one minute after delivery by cesarean section, receiving extra-uterine placental transfusion and physiology-based cord clamping
  Interventions: Procedure: Extrauterine placental transfusion and physiology-based umbilical cord clamping
- Infants with respiratory support: Infants with no or poor spontaneous onset of respiration after delivery by cesarean section, receiving extra-uterine placental transfusion, intact-cord stabilisation (any respiratory support) and physiology-based cord clamping after transfer to resuscitation table
  Interventions: Procedure: Extrauterine placental transfusion, intact cord stabilisation and physiology-based umbilical cord clamping
- Historical control group: Infants delivered by cesarean section in a time period when delayed cord clamping after 1-3 minutes was default procedure. Less-than-vigorous infants needing respiratory support or full resuscitation had their umbilical cords cut early (within 30 seconds)
  Interventions: Procedure: Delayed umbilical cord clamping

INTERVENTIONS:
Procedure: Extrauterine placental transfusion and physiology-based umbilical cord clamping — Placenta is delivered prior to umbilical cord clamping to facilitate placental transfusion. Infant and placenta are transferred to a warmer in an adjacent room, the umbilical cord is clamped and cut when the cord is white, pulsations have ceased and the infants is breathing regularly (within 10 minutes after delivery)
  Groups: Self-breathing infants
Procedure: Extrauterine placental transfusion, intact cord stabilisation and physiology-based umbilical cord clamping — Placenta is delivered prior to umbilical cord clamping to facilitate placental transfusion. Infant and placenta are transferred to a warmer in an adjacent room and necessary respiratory support is initiated (CPAP or PPV) by a neonatal team. The umbilical cord is clamped and cut when the cord is white, pulsations have ceased and the infant is breathing regularly with or without support (at maximum 10 minutes after delivery)
  Groups: Infants with respiratory support
Procedure: Delayed umbilical cord clamping — Umbilical cord is clamped and cut minimum 60 seconds after delivery to facilitate placental transfusion. Placenta is delivered after cord clamping. Infants needing respiratory support or other stabilisation are transferred to a warmer in the adjacent room where a neonatal team is waiting.
  Groups: Historical control group

SUMMARY:
This is a feasibility study with historical control designed to evaluate whether delivery of the placenta prior to umbilical cord clamping at caesarean sections is a feasible, safe and acceptable way of facilitating intact-cord stabilisation of preterm and term newborn infants.

DETAILED DESCRIPTION:
Standard procedure when an infant is delivered by caesarean section is to wait to clamp the umbilical cord for approximately one minute, and then transfer the infant to a designated area for assessment and stabilisation. If the infant needs immediate resuscitation, the umbilical cord is cut earlier to expedite transfer to resuscitation equipment and qualified care (including stimulation, clearing airways and respiratory support).

It has been suggested in several pilot and clinical studies that keeping the umbilical cord intact during the infant's transition from intra- to extrauterine life may improve outcomes and survival, especially for preterm infants. Since length of the umbilical cord is limited, finding ways to avoid cutting the cord while initiating stabilisation and care is warranted. To date, most studies have reported on interventions that involve mobile resuscitation equipment; thus keeping the infant in close proximity to the mother. This may be extra challenging in caesareans sections, especially due to space constraints and maintenance of sterility.

The objective of this study to determine whether extra-uterine placental transfusion to facilitate intact-cord stabilisation and physiology-based cord clamping for infants delivered by caesarean section is feasible, safe and acceptable for infants and their mothers, as well as for involved personnel.

ELIGIBILITY:
Inclusion Criteria:

* live infants (singletons or dichorionic twins) born in gestational week 32+0 to 42+0
* delivered by CS in regional anaesthesia
* immediate care may be planned with involved personnel prior to delivery
* informed maternal consent is obtained (parental consent on behalf of the unborn child).

Exclusion Criteria:

* twins, triplets
* significant congenital malformations
* placenta complications with high risk of abnormal maternal blood loss
* severe fetal distress requiring cesarean section in general anaesthesia (crash CS)
* participation in any other clinical study within the last month
* not sufficient time for preparations or collection of maternal/parental consent
* mother does not comprehend Norwegian or English

Ages: 32 Weeks to 42 Weeks | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Women planning to give birth at Clinic Ålesund are candidates for enrolment in this clinical study. Pregnant women will be invited to participate when called for second trimester routine ultrasound scan. They will be asked for preliminary consent in the event of intrapartum or planned cesarean section and fullfilment of inclusion cirteria. Women having ultrasound scans done elsewhere, who are later referred to Clinic Ålesund, may be invited to participate after admission, but will not be approached for consent if delivery is imminent. Both parents (if applicable) must consent on behalf of their infant
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Intervention fidelity (cohort 1) | First 10 minutes after delivery
  Extra-uterine placental transfusion + physiology-based cord clamping applied (for vigorous infants), measured as proportion of completed checklists. Registered by staff, using checklists in the operating room.
Intervention fidelity (cohort 2) | First 10 minutes after delivery
  Extra-uterine placental transfusion + intact-cord stabilisation + physiology-based cord clamping applied (for infants needing any respiratory support), measured as proportion of completed checklists. Registered by staff, using checklists in the operating room.

SECONDARY OUTCOMES:
Dry-electrode ECG attached (cohort 1+2) | Within 10 seconds after birth
  Time from birth to dry-electrode ECG (NeoBeat) is attached to the infant's chest or abdomen (measured in seconds). Registered on a checklist by a time-keeper in the operating room.
First cry or breathing effort (cohort 1+2) | Within 10 minutes after birth
  Time from birth to infant's first cry or attempt of spontaneous breathing (measured in minutes and seconds). Assessed by attending midwife or pediatric registrar. Registered on a checklist by a time-keeper in the operating room.
Heart rate (cohort 1+2) | First 10 -15 minutes after birth
  Infant's heart rate after birth measured by a dry-electrode ECG (NeoBeat). Registered on a special data collection sheet by a timekeeper or attending midwife. Data are transferred wirelessly from the NeoBeat device to the Liveborn App (installed on a designated tablet) for storage and further analysis.
Umbilical cord blood samples (cohort 1+2) | Within 40-60 seconds after birth
  Time from birth to sampling for umbilical cord blood gas analysis (arterial and venous) completed (measured in seconds). Registered on a checklist by a time-keeper in the operating room.
Apgar score (cohort 1+2) | At 1 minute after birth
  Composite of heart rate, breathing effort, skin colour, muscle tone and reflexes (each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Assessed by the attending midwife or pediatric registrar, registered on a special data collection sheet by a timekeeper in the operating room
Delivery of placenta (cohort 1+2) | At 1 minute (+/- 10 seconds) after birth
  Time from birth to delivery of the placenta (measured in minutes ans seconds), registered on checklist by a time-keeper in the operating room
Respiratory support (cohort 2) | First 10-15 minutes after birth
  Type of respiratory support applied. Alternatives are: CPAP (Continuous Positive Airway Pressure) or PPV (Positive Pressure Ventilation) Registered on a special data collection sheet by the attending neonatal team or midwife
Duration of respiratory support (cohort 2) | First 10-15 minutes after birth
  Duration of respiratory support (CPAP or PPV), measured in minutes and seconds. Registered on a special data collection sheet by the attending neonatal team or midwife
Apgar score | At 5 minutes after birth (cohort 1+2)
  Composite of heart rate, breathing effort, skin colour, muscle tone and reflexes (each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Assessed and registered on a special data collection sheet by the attending midwife or neonatal nurse
Stabilisation (cohort 2) | Within 10-20 minutes after birth
  Time from birth to stabilisation achieved (regular breathing, heartrate (HR) >100, Saturation (SpO2) >85%, inspired oxygen fraction (FiO2) <40%. Measured in minutes and seconds. Assessed and registered on a special data collection sheet by the attending midwife or neonatal nurse
Cord clamping time (cohort 1+2) | Within 10 minutes after birth
  Time from birth to umbilical cord clamping (measured in minutes and seconds), registered on a special data collection sheet by the attending midwife
Apgar score (cohort 1+2) | At 10 minutes after birth
  Composite of heart rate, breathing effort, skin colour, muscle tone and reflexes (each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Assessed and registered on a special data collection sheet by the attending midwife or neonatal nurse
Skin-to-skin-contact (cohort 1+2) | Within 2 hours after birth
  Time from birth to continuous skin-to-skin contact between infant and mother (or other parent), measured in minutes. Registered on a checklist by the attending midwife or neonatal nurse
Residual placenta volume (cohort 1+2) | Within 10-15 minutes after birth
  Drained and weighed residual blood volume from placenta and umbilical cord after cord clamping (measured in grams, converted to milliliters by a ratio of 1.05:1). Registered by the attending midwife or assistant nurse

OTHER OUTCOMES:
Post-cesarean infection (all cohorts) | Within14 days after surgery (cesarean section)
  Prevalence of maternal post-operative wound infection needing antibiotic therapy. Registered in a dedicated paper form in the patient's record by the attending obstetrician
Abnormal blood loss (all cohorts) | 45 minutes from incision time
  Prevalence of abnormal maternal blood-loss during surgery and wound closure (more than 1000 ml). Estimated by staff by visual inspection and count of blood-soaked compresses. Registered in the patient's record by the attending obstetrician
Pre-operative maternal Hemoglobin | Within 48 hours before cesarean section
  Maternal Hemoglobin value from a venous blood sample taken before cesarean section, measured in grams per 100 ml. Registered on a checklist and in the patient's record by the midwife
Post-operative maternal Hemoglobin | Within 24 hours after cesarean section
  Maternal Hemoglobin value from a venous blood sample taken after cesarean section, measured in grams per 100 ml. Registered on a checklist and in the patient's record by the midwife
Low Apgar score (all cohorts) | At 5 minutes after birth
  Prevalence of infant Apgar score less than 7 (mild asphyxia), composite of heart rate, breathing effort, skin colour, muscle tone and reflexes (subscale range from 0-2). Assessed and registered on a special data collection sheet and in the patient's record by the attending midwife or neonatal team
Infant hypothermia (all cohorts) | Within 2 hours after birth
  Prevalence of infant rectal temperature less than 36.5 degrees celsius, measured by a thermometer and registered on a special data collection form and in the patient's record by the attending midwife or neonatal team
Admittance to Neonatal Intensive Care Unit (NICU) (all cohorts) | Within 24 hours after birth
  Indication for infant's admittance to neonatal intensive care unit after birth. Assessed by the attending pediatric registrar or neonatologist. Registered in a special data collection sheet and in the patient's record
Days in NICU (all cohorts) | Maximum 2 months
  Infant's length of stay i neonatal intensive care unit, measured in days. Registered on a checklist and in the patient's record by the neonatal team

CONTACTS AND LOCATIONS:
Overall Officials: Beate H Eriksen, MD/PhD, Principal Investigator — Møre and Romsdal Hosptal Trust / Norwegian University of Science and Technology
Locations (1):
- Møre and Romsdal Hospital Trust, Ålesund, Møre and Romsdal, Norway